CLINICAL TRIAL: NCT06312137
Title: A Phase 3 Randomized Open-Label Study of Adjuvant Pembrolizumab With or Without MK-2870 in Participants With Resectable Stage II to IIIB (N2) NSCLC Not Achieving pCR After Receiving Neoadjuvant Pembrolizumab With Platinum-based Doublet Chemotherapy Followed by Surgery
Brief Title: A Study to Assess Efficacy and Safety of Pembrolizumab With or Without Sacituzumab Tirumotecan (MK- 2870) in Adult Participants With Resectable Non Small Cell Lung Cancer (NSCLC) Not Achieving Pathological Complete Response (pCR) (MK-2870-019)
Acronym: TroFuse-019
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2870-019; 2023-508012-35-00 (Registry Identifier: EU CT); MK-2870-019 (Other: MSD); jRCT2021240020 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); U1111-1297-4260 (Other: UTN)
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Carcinoma; Lung cancer; Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma; Lung Neoplasms | interventions — pembrolizumab; Cisplatin; Pemetrexed; Gemcitabine; Carboplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: This is a multi site study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Sacituzumab tirumotecan (Experimental): Participants will receive pembrolizumab 200 mg intravenous (IV) infusion every 3 weeks (Q3W) for up to 12 weeks + double-platinum chemotherapy per neoplasm histology classification at the investigator's discretion as neoadjuvant therapy prior to surgery; followed by sacituzumab tirumotecan 4 mg/kg IV infusion every 2 weeks (Q2W) for up to 12 doses (~24 weeks) with pembrolizumab monotherapy 200 mg IV infusion every 6 weeks (Q6W) for up to 7 cycles (~42 weeks).
  Interventions: Biological: Sacituzumab tirumotecan; Biological: Pembrolizumab; Drug: Rescue medication
- Pembrolizumab (Active Comparator): Participants will receive pembrolizumab 200 mg intravenous (IV) infusion Q3W for up to 12 weeks + double-platinum chemotherapy per neoplasm histology classification at the investigator's discretion as neoadjuvant therapy prior to surgery; followed by pembrolizumab monotherapy 200 mg IV infusion Q6W for up to 7 cycles (~42 weeks).
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Drug: Pemetrexed; Drug: Gemcitabine; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Biological: Sacituzumab tirumotecan — Sacituzumab tirumotecan to be administered as 4mg/kg IV infusion q2w for up to 24 weeks
  Other Names: MK-2870; sac-TMT; SKB264
  Arms: Pembrolizumab + Sacituzumab tirumotecan
Biological: Pembrolizumab — Pembrolizumab to be administered 400mg by IV infusion q6w for up to 42 weeks
  Other Names: MK-3475
Drug: Cisplatin — Cisplatin is administered as 75 mg/m2 IV infusion q3w for up to 12 weeks as background treatment in neoadjuvant phase
  Arms: Pembrolizumab
Drug: Pemetrexed — Pemetrexed will be administered in the neoadjuvant phase as 500 mg/m2 IV infusion q3w for up to 12 weeks as background treatment in participants with nonsquamous NSCLC.
  Arms: Pembrolizumab
Drug: Gemcitabine — Gemcitabine will be administered in the neoadjuvant phase as 1000 mg/m2 or 1250 mg/m2 IV infusion on day 1 and day 8 q3w for up to 24 weeks as background treatment in participants with squamous NSCLC.
  Arms: Pembrolizumab
Drug: Carboplatin — Carboplatin will be administered in the neoadjuvant phase as AUC 5 mg/mL/min or AUC 6 mg/mL/min IV infusion q3w for up to 12 weeks as background treatment.
  Arms: Pembrolizumab
Drug: Paclitaxel — Paclitaxel will be administered in the neoadjuvant phase as 175 mg/m2 or 200 mg/m2 IV infusion q3w for up to 12 weeks as background treatment.
  Arms: Pembrolizumab
Drug: Rescue medication — Participants are allowed to take rescue medication to prevent hypersensitivity and/or infusion reactions as a premedication to study treatment. At the discretion of the investigator, participants are provided with a prescription for rescue medications. Recommended rescue medications are antihistamine, H2 receptor antagonist, acetaminophen or equivalent, dexamethasone or equivalent. A steroid mouthwash (dexamethasone or equivalent) may be given as prophylaxis for stomatitis/oral mucositis.
  Arms: Pembrolizumab + Sacituzumab tirumotecan

SUMMARY:
This study will assess if adding sacituzumab tirumotecan with pembrolizumab after surgery is effective in treating NSCLC for participants not achieving pathological complete response. The primary hypothesis of this study is sacituzumab tirumotecan plus pembrolizumab is superior to pembrolizumab monotherapy with respect to disease free survival (DFS) as assessed by blinded independent central review (BICR).

ELIGIBILITY:
The key inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has histological or cytological confirmation of squamous or nonsquamous non-small cell lung cancer (NSCLC), resectable clinical Stage II, IIIA or IIIB (with nodal involvement [N2]) per AJCC eighth edition guidelines
* Has confirmation that either epidermal growth factor receptor (EGFR)-directed or anaplastic lymphoma kinase (ALK)-directed therapy is not indicated as primary therapy
* Is able to undergo surgery based on opinion of investigator after consultation with surgeon
* Is able to receive neoadjuvant pembrolizumab and platinum-based doublet chemotherapy
* Applies to screening for the adjuvant period only, before randomization: Has not achieved pathological complete response (pCR) at surgery by local review of pathology.
* Applies to screening for the adjuvant period only, before randomization: Tumor tissue sample from surgical resection has been provided for determination of programmed cell death ligand 1 (PD-L1) and trophoblast cell surface antigen 2 (TROP2) status by central vendor before randomization into the adjuvant period
* Applies to screening for the adjuvant period only, before randomization: Confirmed to be disease-free based on re-baseline radiological assessment as documented by contrast enhanced chest/abdomen/pelvis computed tomography (CT) (or magnetic resonance imaging (MRI)) within 28 days before randomization
* Participants who have AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement are eligible
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy (ART)
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load at screening
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at least 4 weeks before the start of study intervention

Exclusion Criteria:

* Has one of the following tumor locations/types:

  * NSCLC involving the superior sulcus
  * Large cell neuro-endocrine cancer (LCNEC)
  * Sarcomatoid tumor
  * Diagnosis of SCLC or, for mixed tumors, presence of small cell elements
* Has Grade ≥2 peripheral neuropathy
* Has history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, uncontrolled symptomatic arrhythmia, prolongation of QT corrected for heart rate by Fridericia's cube root formula (QTcF) interval to >480 ms, and/or other serious cardiovascular and cerebrovascular diseases within the 6 months preceding study intervention
* Has received prior neoadjuvant therapy for their current NSCLC diagnosis
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks before the first dose of study intervention
* Has received prior radiotherapy within 2 weeks of start of study intervention, or radiation-related toxicities, requiring corticosteroids
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study medication
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Is an HIV-infected participant with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has a concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV deoxyribonucleic acid (DNA)) and Hepatitis C virus (defined as anti-HCV antibody (Ab) positive and detectable HCV ribonucleic acid (RNA)) infection
* Has a history of allogeneic tissue/solid organ transplant
* Has not adequately recovered from major surgery or have ongoing surgical complications
* Severe hypersensitivity (≥Grade 3) to study intervention, any of its excipients, and/or to another biologic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2034-02-21 (Estimated); Study Completion 2034-10-23 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) as assessed by Blinded Independent Central Review (BICR) | Up to ~ 93 months
  DFS is defined as the time from randomization to any recurrence (local, locoregional, regional or distant), occurrence of new primary NSCLC, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to ~ 118 months
  OS is defined as the time from randomization to death due to any cause.
Distant metastasis-free survival (DMFS) as assessed by investigator | Up to ~ 118 months
  DMFS is defined as the time from randomization to the first documented distant metastasis or death due to any cause, whichever occurs first. Distant metastasis refers to cancer that has spread from the original (primary) tumor to distant organs or distant lymph nodes.
Disease-Free Survival (DFS) as assessed by investigator | Up to ~ 118 months
  DFS is defined as the time from randomization to any recurrence (local, locoregional, regional or distant), occurrence of new primary NSCLC, or death due to any cause, whichever occurs first.
Lung Cancer Specific Survival (LCSS) | Up to ~ 118 months
  LCSS is defined as the time from randomization to the date of death due to lung cancer.
Number of Participants Who Experience an Adverse Event (AE) | Up to ~ 118 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Number of Participants Who Discontinue Study Intervention Due to AEs | Up to ~ 118 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who discontinue study treatment due to an AE will be presented.
Change from Baseline in Global Health Status/Quality of Life (QoL) score (Quality of Life Questionnaire (QLQ)-C30 Items 29 and 30) | Baseline and up to ~118 months
  The European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) is a psychometrically and clinically validated instrument appropriate for assessing the health-related quality of life (HRQoL) of cancer patients in oncology studies. Each scale or item is scored between 0 and 100, for the global health status or QoL a higher value indicates a better level of function.
Change from Baseline in Physical Functioning Score (QLQ-C30 Items 1 to 5) | Baseline and up to ~118 months
  The EORTC-QLQ is a psychometrically and clinically validated instrument appropriate for assessing the HRQoL of cancer patients in oncology studies. Each scale or item is scored between 0 and 100, for all physical functional scales, a higher value indicates a better level of function.
Change from Baseline in Role Functioning Score (QLQ-C30 Items 6 and 7) | Baseline and up to ~118 months
  The EORTC-QLQ is a psychometrically and clinically validated instrument appropriate for assessing the HRQoL of cancer patients in oncology studies. Each scale or item is scored between 0 and 100, for all role functional scales, a higher value indicates a better level of function.
Change from Baseline in Dyspnea scores (QLQ-C30 Item 8) | Baseline and up to ~118 months
  The EORTC-QLQ is a psychometrically and clinically validated instrument appropriate for assessing the HRQoL of cancer patients in oncology studies. Each scale or item is scored between 0 and 100, for symptom scales such as dyspnea, a higher value indicates increased severity of symptoms.
Change from Baseline in Coughing scores (QLQ-LC24 Items 31 and 52) | Baseline and up to ~118 months
  The lung cancer module of the EORTC, QLQ-LC24 is a revised and updated version of the Lung Cancer Module QLQ-LC13 and is a supplementary lung cancer specific module to be used along with EORTC QLQ C30. The QLQ-LC24 incorporates 4 multi-item scales to assess coughing, shortness of breath, hair problems, and fear of progression, for symptom scales as for cough, a higher value indicates increased severity of symptoms.
Change from Baseline in Chest pain scores (QLQ-LC24 Item 40) | Baseline and up to ~118 months
  The lung cancer module of the EORTC, QLQ-LC24 is a revised and updated version of the Lung Cancer Module QLQ-LC13 and is a supplementary lung cancer specific module to be used along with EORTC QLQ C30. The QLQ-LC24 incorporates 4 multi-item scales to assess coughing, shortness of breath, hair problems, and fear of progression, for symptom scales as for chest pain, a higher value indicates increased severity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (254):
- United States (46):
  - UAMS Winthrop P. Rockefeller Cancer Institute ( Site 0060), Little Rock, Arkansas
  - Highlands Oncology Group-Research Department ( Site 0062), Springdale, Arkansas
  - Beverly Hills Cancer Center ( Site 0070), Beverly Hills, California
  - The Angeles Clinic and Research Institute ( Site 0040), Los Angeles, California
  - The Angeles Clinic and Research Institute- A Cedars-Sinai Affiliate ( Site 0079), Los Angeles, California
  - UCLA Clinical & Translational Research Center (CTRC) ( Site 0033), Los Angeles, California
  - Hoag Memorial Hospital Presbyterian ( Site 0096), Newport Beach, California
  - San Francisco Oncology Associates ( Site 0066), San Francisco, California
  - Stamford Hospital ( Site 0083), Stamford, Connecticut
  - Mayo Clinic in Florida ( Site 0014), Jacksonville, Florida
  - Mount Sinai Cancer Center ( Site 0038), Miami Beach, Florida
  - Mid Florida Hematology and Oncology Center ( Site 0018), Orange City, Florida
  - Emory University School of Medicine-Phase I ( Site 0056), Atlanta, Georgia
  - Northside Hospital ( Site 0055), Atlanta, Georgia
  - Centricity Research Columbus Cancer Center ( Site 0005), Columbus, Georgia
  - Southeastern Regional Medical Center ( Site 0065), Newnan, Georgia
  - Lewis Cancer and Research Pavilion ( Site 0063), Savannah, Georgia
  - Archbold Cancer Center ( Site 0071), Thomasville, Georgia
  - Edward-Elmhurst Healthcare, Elmhurst Hospital-Nancy W. Knowles Cancer Center ( Site 0017), Elmhurst, Illinois
  - Edward-Elmhurst Healthcare, Edward Hospital-Edward Cancer Center ( Site 0078), Naperville, Illinois
  - Parkview Research Center at Parkview Regional Medical Center ( Site 0089), Fort Wayne, Indiana
  - Indiana University Health Arnett Cancer Center ( Site 0076), Lafayette, Indiana
  - Saint Elizabeth Medical Center Edgewood-Cancer Care Center ( Site 0061), Edgewood, Kentucky
  - LSU Health Baton Rouge North Clinic ( Site 4003), Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group-Medical Oncology ( Site 0080), Baton Rouge, Louisiana
  - New England Cancer Specialists ( Site 0095), Westbrook, Maine
  - Allina Health Cancer Institute - Abbott Northwestern Hospital ( Site 0027), Minneapolis, Minnesota
  - Mayo Clinic - Rochester ( Site 0073), Rochester, Minnesota
  - Mercy Research - David C. Pratt Cancer Center ( Site 0006), St Louis, Missouri
  - Renown Regional Medical Center-Renown Health Medical Oncology ( Site 0037), Reno, Nevada
  - Atlantic Health Morristown Medical Center ( Site 0077), Morristown, New Jersey
  - Cayuga Medical Center ( Site 0086), Ithaca, New York
  - Stony Brook University-Cancer Center ( Site 0054), Stony Brook, New York
  - White Plains Hospital ( Site 0091), White Plains, New York
  - Sanford Fargo Medical Center-Roger Maris Cancer Center ( Site 0057), Fargo, North Dakota
  - Hightower Clinical, LLC ( Site 0084), Oklahoma City, Oklahoma
  - Oregon Health and Science University ( Site 0052), Portland, Oregon
  - Penn State Milton S. Hershey Medical Center-Penn State Cancer Institute ( Site 0059), Hershey, Pennsylvania
  - Lancaster General Hospital - Ann B Barshinger Cancer Institute ( Site 0068), Lancaster, Pennsylvania
  - Saint Joseph's Candler Health System ( Site 4010), Bluffton, South Carolina
  - Medical University of South Carolina-Hollings Cancer Center ( Site 0045), Charleston, South Carolina
  - Sanford Cancer Center ( Site 0053), Sioux Falls, South Dakota
  - Avera Cancer Institute- Research ( Site 0090), Sioux Falls, South Dakota
  - University of Tennessee Medical Center Knoxville ( Site 0082), Knoxville, Tennessee
  - Millennium Research & Clinical Development ( Site 0039), Houston, Texas
  - Huntsman Cancer Institute ( Site 0042), Salt Lake City, Utah
- Argentina (7):
  - Hospital Italiano de Buenos Aires-Clinical Oncology ( Site 0213), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Británico de Buenos Aires-Oncology ( Site 0207), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Sanatorio Británico-Clinical Oncology Department ( Site 0206), Rosario, Santa Fe Province
  - Sanatorio Parque ( Site 0205), Rosario, Santa Fe Province
  - Clínica Mayo de Urgencias Médicas Cruz Blanca S.R.L ( Site 0217), San Miguel de Tucumán, Tucumán Province
  - Hospital Aleman-Oncology ( Site 0202), Buenos Aires
  - Hospital Privado Universitario de Córdoba-Hematology and Oncology ( Site 0204), Córdoba
- Australia (3):
  - Westmead Hospital ( Site 0701), Westmead, New South Wales
  - The Prince Charles Hospital ( Site 0700), Brisbane, Queensland
  - Fiona Stanley Hospital-Medical Oncology ( Site 0705), Murdoch, Western Australia
- Austria (4):
  - Medizinische Universitaet Innsbruck-Department for Internal Medicine V ( Site 1403), Innsbruck, Tyrol
  - Ordensklinikum Linz GmbH Elisabethinen-Department of Pneumology ( Site 1402), Linz, Upper Austria
  - Standort Penzing der Klinik Ottakring-Abteilung für Atemwegs-und Lungenkrankheiten ( Site 1401), Vienna
  - Klinik Floridsdorf-Abteilung für Innere Medizin und Pneumologie ( Site 1400), Vienna
- Belgium (3):
  - Antwerp University Hospital-Thoracic Oncology ( Site 1503), Edegem, Antwerpen
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant-Godinne - Site Godi ( Site 1502), Yvoir, Namur
  - VITAZ ( Site 1500), Sint-Niklaas, Oost-Vlaanderen
- Brazil (6):
  - Liga Norte Riograndense Contra o Câncer ( Site 0301), Natal, Rio Grande do Norte
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre ( Site 0303), Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição ( Site 0302), Porto Alegre, Rio Grande do Sul
  - Instituto de Oncologia Saint Gallen ( Site 0319), Santa Cruz do Sul, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos ( Site 0304), Barretos, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto ( Site 0313), São José do Rio Preto, São Paulo
- Canada (4):
  - Centre Intégré de Santé et de Services Sociaux de la Montérégie-Centre ( Site 0100), Greenfield Park, Quebec
  - Centre Hospitalier de l'Université de Montréal ( Site 0104), Montreal, Quebec
  - St. Marys Hospital Center ( Site 0107), Montreal, Quebec
  - McGill University Health Centre ( Site 0105), Montreal, Quebec
- Chile (4):
  - FALP-UIDO ( Site 0401), Providencia, Region M. de Santiago
  - Centro de Estudios Clínicos SAGA-CECSAGA ( Site 0404), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0400), Santiago, Region M. de Santiago
  - ONCOCENTRO APYS-ACEREY ( Site 0410), Viña del Mar, Región de Valparaíso
- China (27):
  - Beijing Cancer hospital-Thoracic Surgery department I ( Site 1301), Beijing, Beijing Municipality
  - Beijing Peking Union Medical College Hospital-Thoracic surgery department ( Site 1302), Beijing, Beijing Municipality
  - Peking University People's Hospital. ( Site 1300), Beijing, Beijing Municipality
  - Fujian Cancer Hospital-oncology department ( Site 1314), Fuzhou, Fujian
  - The First Affiliated Hospital of Guangzhou Medical University-thoracic surgery department ( Site 1320), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital-Thoracic surgery department ( Site 1313), Guangzhou, Guangdong
  - Henan Cancer Hospital-henan cancer hospital ( Site 1316), Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology-Thoracic Surgery ( Site 1306), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 1308), Wuhan, Hubei
  - Xiangya Hospital Central South University-Thoracic surgery ( Site 1311), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 1312), Changsha, Hunan
  - Nanjing First Hospital ( Site 1310), Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University-Thoracic Surgery Department ( Site 1318), Suzhou, Jiangsu
  - The First affiliated hospital of Nanchang University (Xianghu campus) ( Site 1330), Nanchang, Jiangxi
  - The First Hospital of Jilin University ( Site 1324), Changchun, Jilin
  - The Second Affiliated Hospital of Air Force Medical University ( Site 1332), Xi'an, Shaanxi
  - Shandong Cancer Hospital ( Site 1321), Jinan, Shandong
  - Zhongshan Hospital Fudan University ( Site 1325), Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital-Thoracic Surgery department ( Site 1304), Shanghai, Shanghai Municipality
  - Sichuan Cancer hospital. ( Site 1327), Chengdu, Sichuan
  - The Second People's Hospital of Neijiang ( Site 1322), Neijiang, Sichuan
  - Yunnan Province Cancer Hospital ( Site 1315), Kunming, Yunnan
  - The first Affiliated Hospital, Zhejiang University School of-Thoracic Cardiovascular Surgery Ward ( Site 1303), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 1309), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine ( Site 1328), Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province ( Site 1329), Linhai, Zhejiang
  - Ningbo No. 2 Hospital ( Site 1305), Ningbo, Zhejiang
- Czechia (2):
  - Masarykuv onkologicky ustav-Klinika komplexni onkologicke pece ( Site 1600), Brno, Brno-mesto
  - Nemocnice AGEL Ostrava - Vitkovice a.s.-Plicni oddeleni ( Site 1601), Ostrava, Ostrava Mesto
- France (10):
  - CHRU de Brest ( Site 1804), Brest, Finistere
  - CHU de Toulouse - Hopital Larrey-service de pneumologie ( Site 1801), Toulouse, Haute-Garonne
  - CHU Charles Nicolle ( Site 1803), Rouen, Haute-Normandie
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuytren ( Site 1805), Limoges, Haute-Vienne
  - Clinique Teissier Groupe ( Site 1811), Valenciennes, Nord
  - Centre Jean Perrin - Centre Régional de Lutte contre le Cancer d'Auvergne-ONCOLOGY ( Site 1810), Clermont-Ferrand, Puy-de-Dome
  - Hospices Civils de Lyon - Hopital Louis Pradel ( Site 1809), Bron, Rhone
  - HIA Sainte Anne ( Site 1800), Toulon, Var
  - Hôpital Tenon ( Site 1802), Paris
  - Groupe hospitalier Paris saint Joseph. ( Site 1807), Paris, Île-de-France Region
- Germany (12):
  - Klinikum Esslingen-Klinik für Kardiologie und Pneumologie ( Site 1914), Esslingen am Neckar, Baden-Wurttemberg
  - Universitaetsklinikum Regensburg ( Site 1907), Regensburg, Bavaria
  - Lungenklinik Hemer ( Site 1905), Hemer, North Rhine-Westphalia
  - Katholisches Klinikum Koblenz ( Site 1911), Koblenz, Rhineland-Palatinate
  - Universitätsklinikum Leipzig ( Site 1915), Leipzig, Saxony
  - Krankenhaus Martha-Maria Halle-Dölau-Klinik für Innere Medizin II ( Site 1908), Halle, Saxony-Anhalt
  - Zentralklinik Bad Berka-Klinik für Hämatologie und Onkologie ( Site 1902), Bad Berka, Thuringia
  - SRH Wald-Klinikum Gera-Lungenkrebszentrum ( Site 1900), Gera, Thuringia
  - Evangelische Lungenklinik Berlin-Pneumologie ( Site 1904), Berlin
  - Charité Campus Virchow-Klinikum-Department of Infectious Diseases and Pulmonary Medicine ( Site 1903), Berlin
  - Vivantes Hospital Spandau-Klinik für Innere Medizin, Hämatologie, Onkologie und Gastroenterologie- ( Site 1912), Berlin
  - Helios Klinikum Emil von Behring Berlin-Zehlendorf ( Site 1916), Berlin
- Greece (8):
  - UNIVERSITY HOSPITAL OF PATRAS-DIVISION OF ONCOLOGY ( Site 2006), Pátrai, Achaia
  - 251 Hellenic Air Force General Hospital ( Site 2003), Athens, Attica
  - THORACIC GENERAL HOSPITAL OF ATHENS "I SOTIRIA"-3rd Dept of Internal Medicine and Laboratory, Oncol ( Site 2000), Athens, Attica
  - Athens Medical Center ( Site 2005), Athens, Attica
  - Metaxa Cancer Hospital of Piraeus ( Site 2002), Piraeus, Attica
  - University General Hospital of Heraklion-Internal Medicine-Oncology ( Site 2001), Heraklion, Irakleio
  - University General Hospital of Larissa-Oncology Clinic ( Site 2004), Larissa, Thessaly
  - European Interbalkan Medical Center ( Site 2007), Thessaloniki
- Hong Kong (3):
  - Queen Mary Hospital ( Site 3400), Hksar
  - Hong Kong United Oncology Centre ( Site 3403), Kowloon
  - Queen Elizabeth Hospital ( Site 3402), Yau Ma Tei
- Israel (4):
  - Rambam Health Care Campus-Oncology Division ( Site 2203), Haifa
  - Shaare Zedek Medical Center ( Site 2206), Jerusalem
  - Rabin Medical Center ( Site 2204), Petah Tikva
  - Sheba Medical Center ( Site 2200), Ramat Gan
- Italy (14):
  - Humanitas Istituto Clinico Catanese ( Site 2315), Misterbianco, Catania
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori"-Oncologia Medica ( Site 2302), Meldola, Emilia-Romagna
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 2300), Milan, Lombardy
  - San Paolo - ASST SANTI PAOLO E CARLO ( Site 2314), Milan, Lombardy
  - Fondazione IRCCS San Gerardo dei Tintori-Oncologia ( Site 2301), Monza, Lombardy
  - Istituto Nazionale Tumori Regina Elena-Oncologia Medica 2 ( Site 2309), Rome, Roma
  - Azienda Ospedaliera Universitaria Careggi-SOD ONCOLOGIA MEDICA ( Site 2307), Florence, Tuscany
  - Humanitas Gavazzeni-ONCOLOGY ( Site 2310), Bergamo
  - Ospedale San Martino ( Site 2313), Genova
  - Ospedale San Raffaele-Oncologia Medica ( Site 2311), Milan
  - Azienda Ospedaliero Universitaria di Parma-UO Oncologia Medica ( Site 2312), Parma
  - Fondazione IRCCS Policlinico San Matteo-Oncology ( Site 2303), Pavia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -Medical Oncology ( Site 2306), Roma
  - APSS- Presidio Ospedaliero S. Chiara ( Site 2304), Trento
- Japan (19):
  - National Cancer Center Hospital East ( Site 1202), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 1216), Matsuyama, Ehime
  - Hospital of the University of Occupational and Environmental Health, Japan ( Site 1217), Kitakyushu, Fukuoka
  - Kobe City Medical Center General Hospital ( Site 1213), Kobe, Hyōgo
  - St. Marianna University Hospital ( Site 1207), Kawasaki, Kanagawa
  - Kanagawa Cancer Center ( Site 1206), Yokohama, Kanagawa
  - Kansai Medical University Hospital ( Site 1211), Hirakata, Osaka
  - Kindai University Hospital ( Site 1212), Sakai, Osaka
  - Saitama Prefectural Cancer Center ( Site 1201), Kitaadachi-gun, Saitama
  - Juntendo University Hospital ( Site 1204), Bunkyo-ku, Tokyo
  - Tokyo Medical University Hospital ( Site 1203), Shinjuku, Tokyo
  - National Hospital Organization Kyushu Cancer Center ( Site 1218), Fukuoka
  - Fukushima Medical University Hospital ( Site 1200), Fukushima
  - Hiroshima University Hospital ( Site 1215), Hiroshima
  - Niigata Cancer Center Hospital ( Site 1208), Niigata
  - Okayama University Hospital ( Site 1214), Okayama
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute ( Site 1210), Osaka
  - Nippon Medical School Hospital ( Site 1205), Tokyo
  - Yamagata University Hospital ( Site 1219), Yamagata
- Mexico (6):
  - CIO - Centro de Inmuno-Oncología de Occidente ( Site 0506), Guadalajara, Jalisco
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Servicio de Oncología ( Site 0508), Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca ( Site 0509), Oaxaca City, Oaxaca
  - Unidad de Mastologia Avanzada de Chihuahua S.A de C.V ( Site 0504), Chihuahua City
  - Mediadvance Clinical ( Site 0502), Chihuahua City
  - Oaxaca Site Management Organization S.C. ( Site 0507), Oaxaca City
- Netherlands (8):
  - Amphia Ziekenhuis, locatie Breda Molengracht-long oncologie ( Site 3453), Breda, North Brabant
  - Isala, locatie Zwolle-Poli Longziekten ( Site 3454), Zwolle, Overijssel
  - Leids Universitair Medisch Centrum-Longziekten ( Site 3451), Leiden, South Holland
  - Erasmus Medisch Centrum ( Site 3452), Rotterdam, South Holland
  - Meander Medisch Centrum-Researchbureau Longgeneeskunde ( Site 3458), Amersfoort, Utrecht
  - University Medical Center Groningen ( Site 3459), Groningen
  - Martini Ziekenhuis ( Site 3460), Groningen
  - Sint Antonius Ziekenhuis ( Site 3455), Utrecht
- Auckland City Hospital ( Site 0800), Auckland, New Zealand
- Norway (4):
  - Akershus Universitetssykehus ( Site 2501), Lørenskog, Akershus
  - Drammen Sykehus, Vestre Viken HF ( Site 2502), Drammen, Buskerud
  - Sykehuset Innlandet HF Gjøvik ( Site 2503), Gjøvik, Oppland
  - Oslo universitetssykehus HF. Radiumhospitalet ( Site 2504), Oslo
- Peru (5):
  - IPOR Instituto Peruano de Oncología & Radioterapia-Centro de Investigación ( Site 0604), Lima
  - Oncosalud ( Site 0602), Lima
  - INSTITUTO NACIONAL DE ENFERMEDADES NEOPLASICAS-Medical Oncology ( Site 0600), Lima
  - Instituto Neuro Cardiovascular de las Americas ( Site 0607), Lima
  - Hospital Nacional Edgardo Rebagliati Martins-medical oncology ( Site 0603), Lima
- Poland (8):
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii-Oddzial Onkologii Klinicznej z Pododdzialem Dz ( Site 2602), Poznan, Greater Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny nr 4 w Lublinie ( Site 2611), Lublin, Lublin Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier ( Site 2600), Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 2601), Przemyśl, Podkarpackie Voivodeship
  - Bialostockie Centrum Onkologii ( Site 2604), Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne ( Site 2610), Gdansk, Pomeranian Voivodeship
  - Szpital Specjalistyczny w Prabutach Spolka z o.o. ( Site 2613), Prabuty, Pomeranian Voivodeship
  - Warmińsko - Mazurskie Centrum Chorób Płuc w Olsztynie-Oddzial Onkologii z Pododdzialem Chemioterapii ( Site 2606), Olsztyn, Warmian-Masurian Voivodeship
- Portugal (3):
  - UNIDADE LOCAL DE SAUDE DE MATOSINHOS-Serviço de Oncologia ( Site 2705), Matosinhos Municipality, Porto District
  - Instituto Portugês de Oncologia de Coimbra Francisco Gentil-Oncologia Médica ( Site 2704), Coimbra
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE ( Site 2702), Porto
- Romania (8):
  - MEMORIAL HEALTHCARE INTERNATIONAL S.R.L.. ( Site 2803), Bucharest, București
  - Cardiomed SRL Cluj-Napoca-Medical Oncology ( Site 2801), Cluj-Napoca, Cluj
  - SC Radiotherapy Center Cluj SRL-Oncologie Medicala ( Site 2802), Florești, Cluj
  - Centrul de Oncologie Sfantul Nectarie-Medical ( Site 2805), Craiova, Dolj
  - Spitalul Clinic Municipal De Urgenta Timisoara ( Site 2806), Timișoara, Timiș County
  - SC ONCO CARD SRL ( Site 2808), Brasov
  - Spitalul Clinic De Urgenta Prof Dr Agrippa Ionescu ( Site 2804), Bucharest
  - Institutul Regional de Oncologie ( Site 2807), Iași
- South Korea (7):
  - National Cancer Center-Lung Cancer Center ( Site 1002), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital-Medical Oncology ( Site 1003), Seongnam, Kyonggi-do
  - The Catholic University Of Korea St. Vincent's Hospital-Medical Oncology ( Site 1001), Suwon, Kyonggi-do
  - Chungbuk National University Hospital-Internal medicine ( Site 1000), Cheongju-si, North Chungcheong
  - Keimyung University Dongsan Hospital CRC room 1 ( Site 1006), Daegu, Taegu-Kwangyokshi
  - Asan Medical Center-Lung Cancer Center ( Site 1005), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 1004), Seoul
- Spain (6):
  - Institut Català d'Oncologia - L'Hospitalet-Medical Oncology ( Site 2901), L'Hospitalet de Llobregat, Barcelona
  - CHUS - Hospital Clinico Universitario-Servicio de Oncologia ( Site 2905), Santiago de Compostela, La Coruna
  - Hospital Insular de Gran Canaria-Oncology ( Site 2903), Las Palmas de Gran Canaria, Las Palmas
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID-ONCOLOGIA MEDICA ( Site 2902), Pozuelo de Alarcón, Madrid
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 2900), Barcelona
  - Hospital Clinico San Carlos-Oncology Department ( Site 2904), Madrid
- Switzerland (4):
  - CHUV (centre hospitalier universitaire vaudois) ( Site 3003), Lausanne, Canton of Vaud
  - Kantonsspital Graubünden-Medizin ( Site 3006), Chur, Kanton Graubünden
  - Kantonsspital Münsterlingen - Spital Thurgau AG ( Site 3005), Münsterlingen, Thurgau
  - HFR Fribourg - Hôpital Cantonal ( Site 3004), Fribourg
- Taiwan (7):
  - National Taiwan University Cancer Center (NTUCC) ( Site 1105), Taipei City, Taipei
  - Tri-Service General Hospital ( Site 1100), Taipei City, Taipei
  - Taoyuan General Hospital ( Site 1106), Taoyuan, Taoyuan
  - Kaohsiung Medical University Chung-Ho Memorial Hospital ( Site 1103), Kaohsiung City
  - Taichung Veterans General Hospital-Chest ( Site 1101), Taichung
  - National Cheng Kung University Hospital-Clinical Trial Center ( Site 1102), Tainan
  - National Taiwan University Hospital-Oncology ( Site 1104), Taipei
- Turkey (Türkiye) (6):
  - Adana Medical Park Seyhan Hastanesi-Medikal Onkoloji ( Site 3106), Adana
  - Gulhane Egitim Arastirma Hastanesi-Onkoloji ( Site 3104), Ankara
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 3101), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 3110), Ankara
  - Ankara Bilkent Şehir Hastanesi-Medical Oncology ( Site 3103), Ankara
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 3107), Istanbul
- United Kingdom (5):
  - Addenbrooke's Hospital ( Site 3217), Cambridge, Cambridgeshire
  - Mount Vernon Hospital ( Site 3218), Northwood, Hillingdon
  - St Bartholomew's Hospital-Centre for Experimental Cancer Medicine ( Site 3203), London, London, City of
  - Churchill Hospital ( Site 3219), Oxford, Oxfordshire
  - Freeman Hospital-Northern Centre for Cancer Care ( Site 3212), Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26289&tenant=MT_MSD_9011